CLINICAL TRIAL: NCT05630365
Title: Clinical Evaluation of the Panbio™ COVID-19/Flu A&B Rapid Panel Professional Use Product Using Mid-Turbinate Nasal Swabs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Rapid Dx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SDRD-H-027-P
Record Dates: First submitted 2022-11-22; First posted 2022-11-29 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: COVID-19; Influenza A; Influenza Type B
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nasal sampling/Testing (Professional Use) (Experimental): operators will collect one mid-turbinate nasal swab sample from both nostrils from each subject. The collected mid-turbinate nasal swab will be tested with the Panbio™ Rapid Panel by an operator at the study site in a Near Patient Testing setting (e.g. GP centre or hospital clinic). After the mid-turbinate nasal sampling, the operators will collect one NP swab sample from one nostril of each subject.UTM samples will be shipped to the Core Laboratory for testing with RT-PCR protocols for Flu A, Flu B and SARS-CoV-2, as per the laboratory manual
  Interventions: Diagnostic Test: Panbio™

INTERVENTIONS:
Diagnostic Test: Panbio™ — The Panbio™ COVID-19/Flu A&B Rapid Panel device, hereafter referred to as the Panbio™ Rapid Panel, is a visual lateral flow assay for the rapid immuno-chromatographic qualitative detection of COVID-19 antigen, Influenza A antigen, and Influenza B antigen in mid-turbinate nasal swabs
  Other Names: Panbio™ COVID-19/Flu A&B Rapid Panel Professional Use Product

SUMMARY:
This study is designed as an international, prospective, multicentric, clinical study to investigate the performance of the Panbio™ COVID-19/Flu A&B Rapid Panel for the qualitative detection of COVID-19 antigen, Influenza A antigen, and Influenza B antigen in human mid-turbinate nasal swabs collected by a trained health worker. This study is part of the performance evaluation to support the CE conformity assessment procedures.

DETAILED DESCRIPTION:
A minimum of 1531 male and female subjects will be prospectively enrolled at multiple clinical sites to assess the performance of the Panbio™ Rapid Panel in detecting predominant Covid-19 and Flu variants currently in global circulation. A minimum of 120 Flu A reference positive subjects, a minimum of 120 Flu B reference positive subjects and a minimum of 300 SARS-CoV-2 reference positive subjects will be enrolled. In addition, a minimum of 991 reference negative subjects will be enrolled.

After informed consent has been obtained, operators will collect one mid-turbinate nasal swab sample from both nostrils from each subject. The nasal collection procedure will be a mid-turbinate nasal swab (deep nasal swab), by turning the swab five times in each nostril. Mid-turbinate nasal samples must be collected prior to the NP sampling. The collected mid-turbinate nasal swab will be tested with the Panbio™ Rapid Panel by an operator at the study site in a Near Patient Testing setting (e.g. GP centre or hospital clinic).

After the mid-turbinate nasal sampling, the operators will collect one NP swab sample from one nostril of each subject. NP sampling should be performed by trained healthcare professionals who routinely conduct NP sampling as part of their other standard of care and clinical duties. The collected NP swab will be eluted in UTM, provided by Abbott/the Core Laboratory, labelled and stored, according to the laboratory manual. UTM samples will be shipped to the Core Laboratory for testing with RT-PCR protocols for Flu A, Flu B and SARS-CoV-2, as per the laboratory manual. The RT-PCR methods used by the Core Laboratory will be CE marked and FDA cleared, with COVID-19 and Flu assay clearance for NP specimens. Leftover UTM from running RT-PCR should be labelled with subject ID and frozen at -80oC.Discordant results will be investigated as outlined in the laboratory manual.

All other aspects of the subject's care will remain the same with no deviation from prescribed practice. If additional Nasal/NP sampling is required, this must be done after the study procedures outlined in this clinical protocol.

Each operator who performs a Panbio™ COVID-19/Flu A&B Rapid Panel test will fill out a user evaluation questionnaire once, to assess the usability of the device.

Each subject's demographic information, symptomology data, and professionally performed test result and questionnaire will be recorded on source documentation and transferred to an Electronic Data Capture system.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from all age groups, able and willing to provide written informed consent or assent, suspected of having a respiratory viral infection consistent with COVID-19 and or Flu by their healthcare provider within the first five days of the onset of symptoms, and presenting at least two of the following symptoms: fever, headache, tiredness, dry cough, sore throat, runny or stuffy nose, muscle aches, loss of smell, loss of taste or shortness of breath, will be prospectively enrolled.

Exclusion Criteria:

* Subject has had a nasal or a NP swab taken within the last 4 hours and is not available for further testing after 4 hours has elapsed.
* Subject has active nose bleeds or acute facial injuries/trauma.
* Subject has received a nasal vaccine (i.e., FluMist®) within the previous fourteen (14) days.
* Subject is currently taking or has taken an antiviral medication-e.g., Amantadine, Rimantadine, Relenza® (Zanamivir), Tamiflu® (Oseltamivir Phosphate), and Flumadine®-for influenza or COVID-19 within the previous thirty (30) days.
* Subject is currently enrolled in a study to evaluate an investigational drug.
* Subject is unwilling or unable to provide informed consent.
* Vulnerable populations as deemed inappropriate for study by the site's PI and/or reviewing REC.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1129 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Primary Outcome: | immediate
  Evaluate the clinical performance (sensitivity/specificity) of the Panbio™ COVID-19/Flu A&B Rapid Panel in fresh collected mid-turbinate nasal swab specimens from individuals suspected of respiratory viral infection consistent with COVID-19 and/or Flu by their healthcare provider within the first five days of the onset of symptoms in a Near Patient Testing setting, compared to Flu and SARS-CoV-2 RT-PCR tested using NP swab samples. Concordance analyisis of investigational device and reference method. Acceptance criterion: Sensitivity >80%, Specificity >95%

SECONDARY OUTCOMES:
Secondary Outcome: | immediate
  To assess the usability of the Panbio™ Rapid Panel when used by trained healthcare workers using a questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- UCCT @ Complete Health Partners- Nashville, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No